CLINICAL TRIAL: NCT04053595
Title: Estimated Oxygen Extraction Versus Dynamic Parameters for Perioperative Hemodynamic Optimization of Patients Undergoing Non-cardiac Surgery: a Non-inferiority Randomized Controlled Trial
Brief Title: Estimated Oxygen Extraction Versus Dynamic Parameters for Perioperative Hemodynamic Optimization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Abele Donati, MD, Professor, Università Politecnica delle Marche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CLRZ01-19
Record Dates: First submitted 2019-06-11; First posted 2019-08-12 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Perioperative/Postoperative Complications; Morality
Keywords: Peri-operative goal-directed therapy; Hemodynamic optimization; Postoperative complications; Mortality
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Estimated Oxygen Extraction (Experimental)
  Interventions: Diagnostic Test: Estimated oxygen extraction protocol
- Dynamic Parameters (Active Comparator)
  Interventions: Diagnostic Test: Dynamic parameters of fluid responsiveness protocol

INTERVENTIONS:
Diagnostic Test: Dynamic parameters of fluid responsiveness protocol — Dynamic parameter of fluid responsiveness (pulse pressure variation/stroke volume variation) are used to optimize hemodynamics intraoperatively and during the first 6 hours postoperatively when appropriate. A cutoff of 12% is used to predict an increase of stroke volume >10% after fluid administration.
  Arms: Dynamic Parameters
Diagnostic Test: Estimated oxygen extraction protocol — Oxygen extraction is estimated by the difference of arterial oxygen saturation and central venous oxygen saturation divided by arterial oxygen saturation. A cutoff of 27% is used as a marker of inadequate tissue perfusion requiring hemodynamic optimization.
  Arms: Estimated Oxygen Extraction

SUMMARY:
The aim of the study is to evaluate the complications rate of high risk patients undergoing non-cardiac surgery that receive two different protocols of hemodynamic optimization. A group of patients receive a protocol based on dynamic parameters of fluid responsiveness; the other group of patients receive a protocol based of the optimization of oxygen extraction.

The hypothesis is that a perioperative hemodynamic optimization protocol based on oxygen extraction is not inferior to a protocol based on dynamic parameters of fluid responsiveness considering the complication rate developed postoperatively.

DETAILED DESCRIPTION:
Any surgical intervention is a trauma for the organism and a stress response is activated to cope the external insult. This stress response is responsible of an increase in oxygen consumption. If patient is not able to overcome the deficit in oxygen consumption (VO2) during the first hours postoperatively, he/she will go toward complications (in case of delay to meet metabolic demand) or death (in case of persistent VO2 deficit). Therefore, several protocols have been developed to optimise haemodynamic parameters with the aim to reduce tissue hypoperfusion coming from maldistribution or inadequate perfusion and meet the increased metabolic need as soon as possible.

Every patient that probably will not be able to face the surgical stress himself might benefit from modulation of haemodynamic parameters. Actually, goal directed therapy (GDT) is able to improve survival only in high-risk surgical patients. Instead, the reduction of complications rate has been shown also in intermediate-risk population.

Originally, hemodynamic optimisation protocols were developed to reach supranormal value for cardiac output (CO), oxygen delivery (DO2) and VO2. Based on the concept that oxygen extraction rate (O2ER) reflects the balance between DO2 and VO2, a GDT protocol based on O2ER estimation (O2ERe) calculated as (SaO2-ScvO2)/SaO2 has been proposed showing a significantly lower number of organ failure postoperatively compared with control group.

The major determinants of DO2 are cardiac output (CO), haemoglobin level (Hb) and arterial oxygen saturation (SaO2).

An inadequate CO may be optimised using fluids as first line therapy and then inotropes.

In mechanically ventilated patients, heart-lung interaction is useful to recognise in which portion of the Frank-Starling curve the heart of the patient is working and then if CO is able to rise after fluid administration aimed to increase preload. Several parameters based on mini-invasive monitor systems are available to assess fluid responsiveness such as pulse pressure variation (PPV) and stroke volume variation (SVV).

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing general anesthesia and mechanical ventilation for elective major open abdominal surgery (gastrointestinal, urologic, gynecologic and vascular surgery)
* expected duration of surgical procedure higher than 120 minutes
* ASA II-III-IV
* planned postoperative ICU/HDU admission

Exclusion Criteria:

* <18 years old
* pregnancy
* arrhythmia
* arterial curve alteration (resonance, damping) not solvable
* palliative surgical procedures
* denial of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Complications rate | From date of randomization until the date of hospital discharge assessed up to 90 days
  Evaluate the difference of postoperative complications rate between the two groups

SECONDARY OUTCOMES:
Fluid administered | Immediately after the surgery, 6 hours postoperatively and at the date of ICU/HDU discharge assessed up to 90 days
  Evaluate the difference of total amount of fluids administered during the perioperative period between the two groups
Fluid balance | Immediately after the surgery, 6 hours postoperatively and at the date of ICU/HDU discharge assessed up to 90 days
  Evaluate the difference of fluid balance (difference between fluid administered and fluid loss) during postoperative period between the two groups
Vasopressor/inopropic drugs | Immediately after the, 6 hours postoperatively and at the date of ICU/HDU discharge assessed up to 90 days
  Evaluate the difference in needs of vasopressor/inotropic drugs (reporting mean dosage used) between the two groups
Hospital length of stay | From date of randomization until the date of hospital discharge or death from any cause assessed up to 90 days
  Evaluate the difference of total number of days of hospital stay between the two groups
Mortality at day 28 | Day 28 from randomization
  Evaluate the difference of mortality rate at day 28 between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Abele Donati, MD, PhD, Principal Investigator — Università Politecnica delle Marche
Locations (1):
- AOU Ospedali Riuniti Ancona, Ancona, Italy

REFERENCES:
- [Derived] Carsetti A, Amici M, Bernacconi T, Brancaleoni P, Cerutti E, Chiarello M, Cingolani D, Cola L, Corsi D, Forlini G, Giampieri M, Iuorio S, Principi T, Tappata G, Tempesta M, Adrario E, Donati A. Estimated oxygen extraction versus dynamic parameters of fluid-responsiveness for perioperative hemodynamic optimization of patients undergoing non-cardiac surgery: a non-inferiority randomized controlled trial. BMC Anesthesiol. 2020 Apr 18;20(1):87. doi: 10.1186/s12871-020-01011-z. PMID 32305061